CLINICAL TRIAL: NCT00051480
Title: A Single Arm, Phase II Study of TNFerade™ Biologic Gene Therapy + Radiation + 5-FU and Cisplatin in Locally Advanced, Resectable, Esophageal Cancer
Brief Title: Study of TNFerade™ Gene Therapy, Radiation, 5-FU and Cisplatin in Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Purpose: Treatment
Other Study IDs: GV-001.005
Record Dates: First submitted 2003-01-10; First posted 2003-01-13 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

INTERVENTIONS:
Genetic: TNFerade

SUMMARY:
The primary purpose of this study is to assess the safety and feasibility of giving TNFerade™ with 5-FU, Cisplatin and radiation therapy to patients with locally advanced, esophageal cancer prior to surgical resection. TNFerade™ is a replication deficient (E1, E3 and E4 deleted) adenovirus vector containing the gene for TNF-alpha controlled by a radiation inducible promoter. This allows the expression of TNF-alpha to be greatest in the area receiving radiation. TNF-alpha is a potent cytokine that has been shown to have potent anti-cancer activities but, due to systemic toxicity, could not be delivered at effective doses. TNFerade™ is a novel way of selective delivery of TNF-alpha to tumor cells.

TNFerade™ will be delivered once a week for five weeks by direct intratumoral injection by using endoscopy or Endoscopic Ultrasound. 5-FU (1000 mg/m2/day) will be delivered via continuous infusion for 96 hours during weeks 1 and 4. Cisplatin (75 mg/m2) will be delivered on Day 1 and Day 29 intravenously. The dose of radiation delivered will be 45 Gy in 1.8 Gy fractions for 5 weeks.

ELIGIBILITY:
Inclusion criteria:

* 18-75 years for age;
* Patients with biopsy proven locally advanced adenocarcinoma or squamous cell carcinoma of the esophagus, stage II, III, who have not received previous treatment and are considered to have resectable carcinoma;
* Informed consent;
* Karnofsky performance status ≥ 70%;
* Life expectancy greater than 6 months.

Exclusion criteria:

* Diagnosis of lymphoma of the esophagus;
* History of other malignancy in the past 2 years except carcinoma in situ of the cervix or bladder, non-melanomatous skin cancer or localized early stage prostate cancer with patients continuously disease-free;
* Previous chemotherapy or radiation for esophageal cancer or previous radiation therapy to the target field;
* T4 disease, metastatic (stage IV) disease or confirmed invasion of the bronchial tree;
* Extension beyond 2 cm into stomach;
* Liver enzymes >2.0 x ULN (ALT, AST, bilirubin, alkaline phosphatase);
* Coagulopathy (INR >1.5, PTT ratio >1.5);
* Renal insufficiency (creatinine >2.0 mg/dL; calculated creatinine clearance <50 ml/min);
* Significant anemia (hematocrit <28% or hemoglobin <9 g/dL) (may have RBC transfusion), or thrombocytopenia (platelet count <100,000/μL)l or leukopenia (WBC <3,000/µL; ANC <1,500 μL);
* Contraindication to endoscopic or EUS-guided delivery including obstructive lesions that can not be dilated to pass endoscope;
* Clinical evidence of active infection of any type, including hepatitis B or C virus;
* Due to the embryotoxic effects of chemotherapy, pregnant or lactating women, or men unable or unwilling to practice contraception are excluded;
* Experimental medications within the last four weeks prior to Day 1;
* Chronic systemic corticosteriod use (orally or parenterally administered);
* Significant concurrent medical or psychiatric illness as defined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - UCSD Cancer Center, La Jolla, California
  - University of California, Irvine, Orange, California
  - Palo Alto VA Health Care Systems, Palo Alto, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - University Hospitals of Cleveland, Cleveland, Ohio
  - US Oncology, Mary Crowley Center, Dallas, Texas
  - University of Texas/MD Anderson, Houston, Texas
  - Scott & White Center for Cancer Prevention and Care, Temple, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Medical College of Virginia, Richmond, Virginia

REFERENCES:
- [Derived] Chang KJ, Reid T, Senzer N, Swisher S, Pinto H, Hanna N, Chak A, Soetikno R. Phase I evaluation of TNFerade biologic plus chemoradiotherapy before esophagectomy for locally advanced resectable esophageal cancer. Gastrointest Endosc. 2012 Jun;75(6):1139-46.e2. doi: 10.1016/j.gie.2012.01.042. Epub 2012 Apr 18. PMID 22520270